CLINICAL TRIAL: NCT04676841
Title: Assessment of Relationships Between Airborne Microorganisms and Wound Contamination During Orthopaedic Surgery - a Trial Within the Clean Care Project
Brief Title: Wound Contamination During Orthopaedic Surgery
Acronym: Clean Care
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Vastra Gotaland Region (Other Government)
Collaborators: Research Institutes of Sweden (Other); Göteborg University (Other); CRC Medical AB (Unknown); Getinge AB (Unknown); Toul Meditech AB (Unknown); Halmstad University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019-02180
Record Dates: First submitted 2020-11-17; First posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-11

CONDITIONS: Surgical Site Infection; Hip Fractures; Orthopedic Disorder; Implant Infection
Keywords: LAF; UDF; SSI; Wound contamination; Infection control; Airborne contamination; Operating room
MeSH Terms: conditions — Surgical Wound Infection; Hip Fractures; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Swab samples for microbial analysis. Samples taken from skin before surgery and from surgical wound before closure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemiarthroplasty: Hip fracture patients operated with hemiarthroplasty
  Interventions: Device: Conventional ventilation + instrumental tables with integrated laminar airflow; Device: Conventional ventilation + standard instrumental tables; Device: Laminar airflow ventilation + standard instrumental tables

INTERVENTIONS:
Device: Conventional ventilation + instrumental tables with integrated laminar airflow — Surgical instruments protected from contamination by local laminar airflow
Device: Conventional ventilation + standard instrumental tables — Control
Device: Laminar airflow ventilation + standard instrumental tables — Control

SUMMARY:
In the present study we will compare bacteriological findings and the incidence of SSI in relation to laminar airflow (LAF) ventilated ORs, conventional (also called displacement or mixed) ventilated ORs and conventional ventilated ORs with the addition of tables equipped with units providing a local LAF over the surgical instruments.

The hypothesis is that there exist a correlation between number and types of airborne bacteria and bacteria in the surgical wound and on surgical instruments at the time of wound closure.

DETAILED DESCRIPTION:
The scientific literature on the relationship between airborne bacteria and wound contamination during different conditions is scares. A study from 1982 (Whyet et al.), demonstrated that the most important and consistent source of contamination of the wound during clean surgery (in this case hip implant surgery) was via air. The study concluded that approximately one third of bacteria in the wound were caused by direct air contamination whereas the remaining number of bacteria were transferred to the wound by indirect routes such as via contaminated instruments.

The present study includes patients undergoing hemiarthroplastic surgery due to hip fracture.

During the surgery active air sampling, for microbial analysis, will be done within 30 cm from the wound.

Passive sampling of instrument tables, to measure number of depositing bacteria on the surface during the procedure, will be performed by placing sterile filters on the table surfaces before initiating the surgical procedure and collecting them at the end.

Skin and wound sampling will be performed with sterile flocked nylon swabs. The method for skin and wound sampling was decided based on a literature review and discussions with the department of Clinical microbiology at Sahlgrenska University hospital. Both aerobe and anaerobe bacteria will be analyzed.

The wound will be measured and number of personnel, door openings and clothing, at each procedure will be recorded.

Patients included in the study will be interviewed after 6 weeks and 1 year, to evaluate incidence rate of SSI.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing hip fracture surgery treated with hemiarthroplasty implant and that are subsequently cared for at participating ortho-geriatric unit

Exclusion Criteria:

* Patients that will not give their informed consent.
* Patient that, at the time of surgery, have an infection in any part of the body, hospital or community acquired.
* Patients receiving fracture fixation with pins only

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hip fracture patients operated with hemiarthroplasty
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Live bacterial Count (colony forming units, CFU) per meter3 air during surgery; in ORs with LAF ventilation, Conventional ventilation or Conventional ventilation + local LAF above instrument tables | 2019-2021
  Active airsampling within 30cm from the surgical wound will be performed during surgery and number of collected aerobe and anaerobe bacteria analyzed.
Number of CFU in the surgical wound before closure; after surgery in ORs with LAF ventilation, Conventional ventilation or Conventional ventilation + local LAF above instrument tables | 2019-2021
  The entire wound is swabed before closure, aerobe and anaerobe bacteria analyzed.

SECONDARY OUTCOMES:
CFU/dm2 on the patients skin Before directly prior to incission, before surgery in surgery in ORs with LAF ventilation, Conventional ventilation or Conventional ventilation + local LAF above instrument tables | 2019-2022
  Swab sample is taken of the skin directly prior to incission, aerobe and anaerobe bacteria analyzed.
CFU/dm2 on the instrument tables during surgery in ORs with LAF ventilation, Conventional ventilation or Conventional ventilation + local LAF above instrument tables | 2019-2022
  Passive sampling of bacteria falling down on the instrument tables during the duration of each surgical procedure will be analyzed. Aerobe and anaerobe bacteria analyzed.
Bacterial species in air collected during surgery in ORs with LAF ventilation, Conventional ventilation or Conventional ventilation + local LAF above instrument tables | 2019-2022
  The bacterial species in collected samples are identified with MALDI-TOF
Bacterial species in wound samples collected during surgery in ORs with LAF ventilation, Conventional ventilation or Conventional ventilation + local LAF above instrument tables | 2019-2022
  The bacterial species in collected samples are identified with MALDI-TOF
Number and sort of SSI in patients operated in ORs with LAF ventilation, Conventional ventilation or Conventional ventilation + local LAF above instrument tables | 2019-2022
  Patients are contacted 6 weeks and 1 year after surgery and incidense and severrensess of infection recorded

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Malchau, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Department of Ortopedics, Sahlgrenska University Hospital, Mölndal, Sweden